CLINICAL TRIAL: NCT00238784
Title: A Comparison of Symbicort® Single Inhaler Therapy (Symbicort® 200 Turbuhaler® 1 Inhalation b.i.d. Plus as Needed) & Conventional Best Practice for the Treatment of Persistent Asthma in Adolescents & Adults-a 26-Week, Randomised, Open-Label, Parallel Group, Multicentre Study
Brief Title: SOLO-Symbicort® in the Treatment of Persistent Asthma in Adolescents & Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00004; SOLO
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide/formoterol Turbuhaler

SUMMARY:
The purpose of this study is to compare Symbicort Single Inhaler treatment with the Best Conventional Practice in patients with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma < 3 months
* Prescribed daily use of glucocorticosteroids for at least 3 months prior to Visit 1

Exclusion Criteria:

* Smoking history > 10 pack-years
* Asthma exacerbation requiring change in asthma treatment during the last 14 days prior to inclusion
* Any significant disease or disorder that my jeopardize the safety of the patient.

Additional inclusion and exclusion criteria will be evaluated by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of asthma exacerbations
Mean use of as-needed medication
Prescribed asthma medication
Patient reported Outcomes
Health care resource use
Safety: Adverse Events, Serious Adverse Events and discontinuations due to Adverse Events
Induced sputum will be sampled from a subset of patients
All variables assessed over the 6 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Rita Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- Canada (3):
  - Research Site, Aldergrove, British Columbia
  - Research Site, Bolton, Ontario
  - Research Site, Brampton, Ontario

REFERENCES:
- [Derived] Sears MR, Boulet LP, Laviolette M, Fitzgerald JM, Bai TR, Kaplan A, Smiljanic-Georgijev N, Lee JS. Budesonide/formoterol maintenance and reliever therapy: impact on airway inflammation in asthma. Eur Respir J. 2008 May;31(5):982-9. doi: 10.1183/09031936.00104007. Epub 2008 Jan 23. PMID 18216054